CLINICAL TRIAL: NCT00477646
Title: New York Prevention Care Manager Project / Medicaid Managed Care Organization Version
Brief Title: Helping Women Stay Up-To-Date With Cancer Screening By Using a Prevention Care Manager or Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Clinical Directors Network (Network)
Responsible Party: Allen J. Dietrich, MD, Dartmouth Medical School, Department of Community & Family Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR0000537346; P30CA023108 (NIH); DMS-20253
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer; Cervical Cancer; Colorectal Cancer
Keywords: colon cancer; rectal cancer; breast cancer; cervical cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention Care Management (Experimental): Telephone support over 18 months from trained Prevention Care Managers, to help women overcome barriers to colon, breast, and cervical cancer screening
  Interventions: Behavioral: Prevention Care Management
- Usual Care (No Intervention): Usual Care. A sample of patients receive a single telephone call to validate claims data and collect basic demographic information.

INTERVENTIONS:
Behavioral: Prevention Care Management — Telephone support over 18 months to help women become screened for breast, cervical and colon cancer. Includes barriers assessment, patient education and motivation, provider recommendation letter, appointment reminder, and some scheduling of appointments.
  Arms: Prevention Care Management

SUMMARY:
RATIONALE: Women may stay up-to-date with cancer screening if a health professional helps them overcome barriers to screening, including helping them to schedule cancer screening appointments.

PURPOSE: This randomized clinical trial is studying the use of health professional-tailored telephone support compared with usual care from their personal doctor to help women overcome barriers to screening for colorectal, cervical, and breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Develop and evaluate an enhanced telephone support intervention (Prevention Care Manager [PCM]) to promote colorectal, cervical, and breast cancer screening more widely among women enrolled in a Medicaid Managed Care Organization (MMCO).
* Explore the impact of patient, Community/Migrant Health Center (C/MHC), and MMCO characteristics on cancer screening status and the impact of the intervention.
* Evaluate the impact of the enhanced PCM intervention upon colorectal, breast, and cervical cancer screening rates.

Secondary

* Compare the status of women who are up-to-date (UTD) on CRC screening versus the UTD status of cervical cancer and breast cancer screening.

OUTLINE: This is a randomized, controlled study. The study is conducted in 2 parts.

* Part 1 (barrier interview and pilot testing): Patients are stratified according to primary language and whether or not they have had an outpatient visit in the past year.

  * Barrier interview: Patients undergo a 15-30 minute interview to determine barriers they face preventing them from receiving recommended cancer screenings and healthcare, as well as facilitators which have encouraged them to be screened.
  * Pilot testing: Patients from the barrier interviews and other eligible Medicaid Managed Care Organization (MMCO) patients receive scripted telephone calls from a Prevention Care Manager to assist them in getting up-to-date on their cancer screening tests over 3 months.
* Part 2 (randomized control trial): Patients are stratified according to treatment center (Community/Migrant health center vs Diagnostic and Treatment Center) and age. Patient are randomized to 1 of 2 intervention arms.

  * Arm I (Prevention Care Manager): Patients are stratified according to the number of tests for which they are up-to-date at baseline. Patients receive reminder letters encouraging them to contact their primary care provider for colorectal, breast, and cervical cancer screening and 3 to 4 telephone support calls to help them become up to date for colorectal, breast, and cervical cancer screening.
  * Arm II (usual care): Patients receive usual care according to their primary care physician.

In both arms, patients are followed for 18 months.

PROJECTED ACCRUAL: A total of 2,600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled in a participating Medicaid Managed Care Organization (MMCO) as a Medicaid patient for ≥ 12 months
* Not up-to-date (UTD) for colorectal cancer screening

  * UTD status defined by any of the following:

    * Home fecal occult blood test within the past 12 months
    * Flexible sigmoidoscopy within the past 5 years
    * Double-contrast barium enema within the past 5 years
    * Colonoscopy within the past 10 years
* Registered to receive primary care from a participating Community/Migrant Health Center, Diagnostic and Treatment Center, or other participating practice in New York City
* Must have a telephone available
* No MMCO claim for any of the following:

  * Colorectal, breast, or cervical cancer
  * Colon polyp removal
  * Total colectomy

PATIENT CHARACTERISTICS:

* Female
* Able to use telephone
* No plans to move for ≥ 1 year

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2241 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients up-to-date (UTD) for colorectal cancer (CRC) screening | 18 months
  Comparison of women in PCM and UC arms who received colon cancer screening tests during 18 month intervention period.

SECONDARY OUTCOMES:
Percentage of patients UTD for breast and cervical cancer screening | 18 months
Comparison of UTD status for CRC screening with UTD status for cervical cancer and breast cancer screening | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Allen J. Dietrich, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Clinical Directors Network, Incorporated, New York, New York, United States

REFERENCES:
- [Derived] Dietrich AJ, Tobin JN, Robinson CM, Cassells A, Greene MA, Dunn VH, Falkenstern KM, De Leon R, Beach ML. Telephone outreach to increase colon cancer screening in medicaid managed care organizations: a randomized controlled trial. Ann Fam Med. 2013 Jul-Aug;11(4):335-43. doi: 10.1370/afm.1469. PMID 23835819